CLINICAL TRIAL: NCT00432445
Title: A Phase II Trial of Proton Beam Radiation Therapy for Intra- and Periocular Retinoblastoma
Brief Title: Proton Beam Radiation Therapy for Intraocular and Periocular Retinoblastoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0883; NCI-2012-01427 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-02-05; First posted 2007-02-07 (Estimated); Results first posted 2015-02-27 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Retinoblastoma
Keywords: Children with retinoblastoma; Retinoblastoma; Pediatrics; Proton Beam Radiation Therapy; Radiation Therapy; Tumor of the Eye; Ophthalmic EUA; Examination under anesthesia; Bilateral retinoblastoma; Unilateral retinoblastoma; Extraocular disease; Intraocular procedure
MeSH Terms: conditions — Retinoblastoma; Eye Neoplasms | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Proton Beam Radiation Therapy (Experimental): Radiation given daily for 5 days in a row each week (except for Saturdays, Sundays, and holidays). The whole treatment will take about 4-6 weeks. Ophthalmic examination under anesthesia including dilated eye exam, ocular fundus photography (Ret-Cam), ocular echography and neuro-radiologic assessment (as deemed necessary)
  Interventions: Radiation: Proton Beam Radiation Therapy; Procedure: Ophthalmic EUA

INTERVENTIONS:
Radiation: Proton Beam Radiation Therapy — Radiation given daily for 5 days in a row each week (except for Saturdays, Sundays, and holidays). The whole treatment will take about 4-6 weeks.
Procedure: Ophthalmic EUA — Ophthalmic examination under anesthesia including dilated eye exam, ocular fundus photography (Ret-Cam), ocular echography and neuro-radiologic assessment (as deemed necessary)
  Other Names: eye exam; ophthalmic exam

SUMMARY:
The purpose of this trial is to evaluate proton beam radiation therapy as an alternative to external photon beam irradiation in children with retinoblastoma as a means of local tumor control and ocular retention.

DETAILED DESCRIPTION:
External photon beam radiation therapy (which is current standard of care) has been used in the treatment of retinoblastoma. It is a form of radiation therapy in which the radiation is delivered by a machine pointed at the area to be radiated.

Proton beam radiation therapy is a form of external photon beam radiation therapy, but it may be more effective because its adjusted dosing delivers less radiation to surrounding areas of the tumor, which helps preserve other tissues and cause fewer side effects.

Before you can start treatment on this study, you will have what are called "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. Your eye doctor will perform an assessment of your eye, including an exam while you are under anesthesia. This exam will include a dilated eye exam, photography of your affected eye (by a Ret-Cam), ultrasound of your affected eye, and imaging scans, such as computed tomography (CT) or magnetic resonance imaging (MRI), if the doctor thinks it is necessary. The assessments will be done to check and confirm the status of the disease.

After diagnosis of retinoblastoma, the study doctor will first see if external photon beam radiation therapy is a reasonable treatment option for you. If external photon beam radiotherapy is deemed appropriate for you, you will be eligible to receive proton beam radiation therapy in this study.

If you are found to be eligible to take part in this study, you will be treated with proton beam radiation therapy. Treatment will begin within 1 week of referral to the M. D. Anderson Proton Center. It will be given daily for 5 days in a row each week (except for Saturdays, Sundays, and holidays). The whole treatment will take about 4-6 weeks.

Within 2-4 weeks after completion of therapy, you will have an eye exam performed under anesthesia (like the one during screening). You will have repeated eye exams under anesthesia, depending on the appearance and response of the tumor to therapy. This will occur about every 1-4 months.

You will continue to have these eye exams until the tumors are considered to be stable or unless your disease gets worse.

If the disease gets worse or you experience any intolerable side effects, you may be taken off treatment.

You will be required to have lifelong eye and medical assessments to continue to monitor you for disease. If no disease is found 5 years after completion of proton beam radiation therapy, you will be considered free of disease. You will then have annual (yearly) eye and pediatric assessment through adulthood.

This is an investigational study. Up to 20 patients will take part in this study. All will be enrolled at M.D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Active or recurrent retinoblastoma patient eligible for treatment of external beam radiation therapy.
2. A parent or guardian who can provide informed consent to a minor or child participant.
3. No concurrent infection.
4. No contraindication for repeated general anesthesia/sedation.

Exclusion Criteria:

1. Inability to return for multiple examinations under anesthesia.
2. Medical contraindication for exams under anesthesia/sedation.
3. Unreliable follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Gombos, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Study closed early due to low accrual, few eligible participants.
Groups:
- Proton Beam Radiation Therapy: Proton Beam Radiation Therapy given daily for 5 days in a row each week where whole treatment takes about 4-6 weeks. Ophthalmic examination under anesthesia including dilated eye exam, ocular fundus photography (Ret-Cam), ocular echography and neuro-radiologic assessment (as deemed necessary).
Period: Overall Study
Arm/Group | Proton Beam Radiation Therapy
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: No analysis performed as a result of small study population.
Arm/Group | Proton Beam Radiation Therapy
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Rate of Local Control in the Globe at 12 Months
Description: Where proton beam radiation therapy used as an alternative to external photon beam irradiation in children with retinoblastoma as a means of local tumor control and ocular retention, local tumor control measured for participants with a globe as tumor regression with ocular retention, and for post enucleation measured as lack of orbital tumor recurrence.
Time Frame: 12 months
Population: No analysis performed. Study did not meet anticipated enrollment.
Arm/Group | Proton Beam Radiation Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Data collected at time point post radiation therapy for retinoblastoma at the following intervals: 3 months (+/- 1 month), 6 months (+/- 1 month), then annually (+/- 1 month) for the first five years. Overall study period: January 2007 to February 2014.
Arm/Group | Proton Beam Radiation Therapy
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proton Beam Radiation Therapy (N=2)
Retinopathy (Eye disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proton Beam Radiation Therapy (N=2)
Post-radiation keratopathy (Eye disorders) | 2 (2)
Retinopathy (Eye disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes